CLINICAL TRIAL: NCT02945722
Title: Study of the Impact of a Targeted Decolonization of S. Aureus Persistent Carriers on the Occurrence of S. Aureus Infections in Hemodialysis Patients
Brief Title: Study of the Impact of a Targeted Decolonization of S. Aureus Persistent Carriers
Acronym: CIBERSTAPH
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of inclusons
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1608170; 2016-004381-25 (EudraCT Number)
Record Dates: First submitted 2016-10-25; First posted 2016-10-26 (Estimated); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Hemodialysis Patients
Keywords: Hemodialysis; S. Aureus; Decolonization; Persistent carriage
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decolonization (Active Comparator): persistent carriers will be decolonized. Decolonization schedule associate the use of mupirocin nasal ointment 3 times a day and chlorhexidine bath once a day for 5 days.
  Interventions: Drug: Decolonization
- No decolonization (Placebo Comparator): HD patients in which decolonization is not performed including impersistent carriers.
  Interventions: Other: No decolonization

INTERVENTIONS:
Drug: Decolonization — Decolonization schedule associate the use of mupirocin nasal ointment 3 times a day and chlorhexidine bath once a day for 5 days. Screening of persistent carriers will be done every 3 months
  Arms: Decolonization
Other: No decolonization — Screening of persistent carriers in this arm will be done every 3 months
  Arms: No decolonization

SUMMARY:
S. aureus nasal carriage is a well-known risk factor for S. aureus infections in hemodialysis (HD) patients. Strains of carriage and infections are the same in >80% of cases We recently shown that persistent carriers of S. aureus, not intermittent ones are at increased risk of staphylococcal infections in HD. Thanks to a new algorithm developped based on one nasal sample the determination of carriage status (persistent, intermittent or non-carriers) among patients is easy. Mupirocin use in HD have been shown to reduce significantly S. aureus infections however, multiples schedules of decolonization have been proposed to all S. aureus carriers. To date, there is no national guideline for decolonization of S. aureus in HD. We showed that only 50% of HD centers in France propose screening and decolonization of S. aureus carriers. The aim of the study is therefore to evaluate the impact of a targeted decolonization of S. aureus persistent carriers using mupirocin nasal ointment and chlorhexidine baths during 5 days on the occurrence of S. aureus infections in HD patients compared to the absence of decolonization using a randomized open study methodology.

DETAILED DESCRIPTION:
Hemodialysis patients will be randomized in 2 arms: one arm where persistent carriers will be decolonized. Decolonization schedule associate the use of mupirocin nasal ointment 3 times a day and chlorhexidine bath once a day for 5 days. Screening of persistent carriers in this arm will be done every 3 months and a new decolonization will be proposed to patients found (again) persistent carriers. Determination of carriage status will be done using one nasal swab by following the algorithm previously described. Bacterial load will be determined by a quantitative S. aureus PCR (Polymerase Chain Reaction) : persistent carriers are the patient with a bacterial load > 103 CFU/mL (Colony Forming Unit) .

The other arm is HD patients in which decolonization is not performed including impersistent carriers.

All infections that occurred in enrolled patients will be counted in both groups

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥ 18 years-old)
* Patient under chronic hemodialysis
* Patent that accepted to participate in the study with a written consent form signed

Exclusion Criteria:

* Patients under peritoneal dialysis
* Patients with an active infection at the time of inclusion
* Patients previously treated by mupirocin and chlorhexidine for decolonization purpose
* Patients that received antimicrobials active on S. aureus during the month before the inclusion
* Patients with allergy to mupirocin or chlorhexidine
* Patients treated by hemodialysis transiently (non-terminal kidney failure)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 434 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2024-10-26 (Actual); Study Completion 2024-10-26 (Actual)

PRIMARY OUTCOMES:
S. aureus infection | 12 months
  Number of S. Aureus define by Centers for Disease Control

SECONDARY OUTCOMES:
endogenous S. aureus infections | 12 months
  same strain of carriage and infection
Bacteremias S. aureus | 12 months
  Impact of Bacteremias S. aureus
strain of S. aureus | 12 months
  Percentage of resistants strains of S. aureus at mupirocin and chlorhexidine
persistents carriers of S. aureus | Months : 3, 6, 9, 12
  Percentage of persistents carriers of S. aureus
intermittents carriers of S. aureus | Months : 3, 6, 9, 12
  Percentage of intermittents carriers of S. aureus
non-carriers carriers of S. aureus | Months : 3, 6, 9, 12
  Percentage of non-carriers carriers of S. aureus
other bacterial infections | 12 months
  Impact of other bacterial infections without S. aureus

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Botelho-Nevers, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (9):
- France (9):
  - CH d'Annecy-Genevois, Annecy
  - CH Emile Roux, Le Puy-en-Velay
  - Aural, Lyon
  - CH St-Joseph St-Luc, Lyon
  - AIDER Santé, Montpellier
  - ARTIC42, Saint-Etienne
  - Chu Saint-Etienne, Saint-Etienne
  - NephroCare, Sainte-Foy-lès-Lyon
  - CH Yssingeaux - Hôpital Local, Yssingeaux

IPD SHARING:
Plan to Share IPD: No